CLINICAL TRIAL: NCT03482479
Title: Low Dose Naltrexone to Improve Physical Health in Patients With Vasculitis
Acronym: LoDoNaVasc
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VCRC5564
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis (EGPA); Churg-Strauss Syndrome (CSS); Giant Cell Arteritis; Granulomatosis With Polyangiitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis
MeSH Terms: conditions — Churg-Strauss Syndrome; Giant Cell Arteritis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone Hydrochloride (Experimental): Naltrexone hydrochloride for oral use, 4.5 mg per capsule, taken once a day for 6 weeks.
  Interventions: Other: Placebo Comparator
- Placebo Comparator (Placebo Comparator): Placebo to match naltrexone for oral use to be taken once a day for 6 weeks.
  Interventions: Drug: Naltrexone Hydrochloride

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — Naltrexone Hydrochloride will be taken daily (dose 4.5 mg) for six weeks
  Arms: Placebo Comparator
Other: Placebo Comparator — A placebo tablet which matches the drug will be taken daily for 6 weeks.
  Arms: Naltrexone Hydrochloride

SUMMARY:
Naltrexone is an FDA approved drug (for alcoholism) that has found widespread use "off-label" to treat pain and improve quality of life at much lower doses than are used for the approved indication. There are a few scientific studies in three conditions (fibromyalgia, Crohn's disease, and multiple sclerosis) that suggest that this drug has benefit and is safe. However, considering the extent of use in other conditions, and uncertainty about the mechanism of action study is needed in a diverse set of diseases, including vasculitis.

The purpose of this clinical trial is to determine if low dose naltrexone is effective in improving health-related quality of life (HRQoL) among patients with vasculitis. Although it is a pilot study, a placebo-controlled component is used because of the prominent placebo group effect seen in studies with self-reported subjective outcomes.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, cross-over, placebo-controlled trial to evaluate the efficacy of low-dose naltrexone (LDN) 4.5 mg nightly in improving self-reported physical health in patients with vasculitis.

At study enrollment, each patient will be randomized to receive either LDN for 6 weeks followed by oral placebo for 6 weeks, or placebo for 6 weeks followed by LDN for 6 weeks. The primary outcome measure and some secondary outcome measures are patient-reported and will be recorded every 3 weeks, or every 6 weeks

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria in order to be eligible for enrollment:

1. Criteria for diagnosis of giant cell arteritis (GCA), Takayasu's arteritis (TAK), polyarteritis nodosa (PAN), granulomatosis with polyangiitis (GPA, Wegener's), microscopic polyangiitis (MPA), or eosinophilic granulomatosis with polyangiitis (EGPA, Churg-Strauss), as used for the VCRC longitudinal studies

a. Giant cell arteritis: According to the American College of Rheumatology (ACR) criteria for classification of GCA, meeting at least 2 of the following 5 remaining criteria at the time of diagnosis of GCA: Age of disease onset >50 years (required) i. New onset or new type of localized pain in the head ii. Temporal artery abnormality (i.e. temporal artery tenderness to palpation or decreased pulsation, unrelated to arteriosclerosis of cervical arteries) iii. ESR of >40 mm in the first hour by Westergren method iv. Temporal artery biopsy showing vasculitis characterized by a predominance of mononuclear cell infiltration or granulomatous inflammation, usually with multinucleated giant cells v. Large Vessel Vasculitis (LVV) by angiogram or biopsy not explained by something else

b. Takayasu's arteritis: According to an adaption of the American College of Rheumatology criteria, meeting at least 2 of the following 5 remaining criteria at the time of inclusion of TAK: Arteriogram abnormalities compatible with TAK (includes conventional dye angiography or MR angiography or CT angiography) (required) i. Age at disease onset ≤50 years ii. Claudication of extremities iii. Decreased brachial artery pulse (one or both arteries) iv. Blood pressure difference of >10mm Hg between the arms v. Bruit over subclavian arteritis or aorta

c. Polyarteritis nodosa: An adaption of the America College of Rheumatology criteria will be used for the diagnosis of PAN. At the time of inclusion, one major and one minor criteria or two major criteria or isolated cutaneous PAN must be met.

i. Major criteria (not explained by other causes):

1. Arteriographic abnormality
2. Presence of granulocyte or mixed leukocyte infiltrate in an arterial wall on biopsy
3. Mononeuropathy or polyneuropathy ii. Minor criteria (not explained by other causes)

1. Weight loss > 4 kg 2. Livedo reticularis, cutaneous ulcerations, or skin nodules 3. Testicular pain or tenderness 4. Myalgias 5. Diastolic blood pressure >90mm Hg 6. Elevated BUN or serum creatinine levels 7. Ischemic abdominal pain iii. Isolated cutaneous polyarteritis nodosa

1. Biopsy-proven cutaneous PAN

   d. Granulomatosis with polyangiitis: Participants can be enrolled if two of the five modified American College of Rheumatology criteria are met: i. Nasal or oral inflammation: painful or painless oral ulcers or purulent or blood nasal discharge ii. Abnormal chest radiograph: nodules, fixed infiltrates, or cavities iii. Urinary sediment: microhematuria or red cell casts iv. Granulomatous inflammation on biopsy: granulomatous inflammation within the wall of an artery or in the perivascular area v. ANCA positivity by enzyme immunoassay for either PR3- or MPO-ANCA e. Microscopic polyangiitis: The following Chapel Hill Consensus Conference Definitions for MPA need to be met: i. Necrotizing vasculitis with few or no immune deposits affects small vessel (i.e., capillaries, venules, or arterioles) ii. Necrotizing arteritis involving small and medium-sized arteritis may be present iii. Necrotizing glomerulonephritis is very common iv. Pulmonary capillaritis often occurs

   f. Eosinophilic granulomatosis with polyangiitis: An adaptation of the American College of Rheumatology criteria will be used for the diagnosis of EGPA. At the time of inclusion, four of the six items must have documented evidence: i. Asthma ii. Peak peripheral blood eosinophilia of >10% of total WBC iii. Peripheral neuropathy attributable to vasculitis iv. Transient pulmonary infiltrates on chest imaging studies v. Paranasal sinus abnormalities or nasal polyposis vi. Eosinophilic inflammation on tissue biopsy If patients have 4 of the above 6 criteria but lack clear-cut documentation of small vessel vasculitis, they are also eligible for enrollment.
2. Baseline normalized score on PROMIS Global Physical Health of 40 or lower.
3. Vasculitis in remission or very low disease activity, as defined by Physician Global Assessment 0-1 for at least 12 weeks
4. Stable immunosuppressive therapy (including prednisone) related to vasculitis for at least 12 weeks
5. No change in medications in the past 12 weeks made with the expectation of improving pain, fatigue, or mood
6. No plan to change medication or a non-pharmacologic treatment regimen likely to affect pain, fatigue, mood, or vasculitis activity during the next 12 weeks
7. Age of 18 years or older
8. Willingness and ability to comply with treatment and follow-up procedures, including receipt of weekly phone calls from the study coordinator
9. Willingness and ability to provide informed consent -

Exclusion Criteria:

1. Change in any medication related to control of vasculitis, pain, fatigue, or mood within the past 12 weeks (medications taken as needed must be in a stable pattern per the patient's estimation)
2. Use of another investigational agent as part of a clinical trial within 30 days of enrollment
3. Current use of any opioid agonist including tramadol or suboxone
4. Change in vasculitis activity in the past 12 weeks, as defined by a change in Physician Global Assessment greater than 1
5. Baseline normalized score more than 40 on PROMIS Global Physical Health
6. New major medical problem or surgery in past 12 weeks
7. Pregnancy or breastfeeding
8. Inability to provide informed consent or comply with study procedures
9. Schizophrenia or bipolar disorder
10. Poorly controlled depression or anxiety, as defined by a score of ≥ 20 on PHQ-9
11. Liver cirrhosis
12. Significant kidney disease, defined as glomerular filtration rate <30ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
PROMIS Global Physical Health | Week 12.
  Questionnaire about improved health related quality of life to a greater extent than placebo.

SECONDARY OUTCOMES:
PROMIS Global Physical Health | 9 weeks
  Questionnaire about improved health related quality of life to a greater extent than placebo.
SF-36 (physical component subscore) | 12 weeks
  Health related quality of life measured by a questionnaire.
PROMIS Questionnaires | 12 weeks
  Questions will ask about anxiety, depression, and sleep disturbance on the PROMIS short form, PROMIS Global Mental Health, and on PROMIS-CAT will ask about physical function, fatigue, satisfaction with social roles, and pain interference, as well in the pain intensity item.
Clinical Global Impression of Severity (CGI-S) | 12 weeks
  7-point scale of patients' self-reporting of severity during the study.
Clinical Global Impression of Improvement (CGI-I) | 12 weeks
  7-point scale of patients' self-reporting of severity during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Merkel, MD, MPH, Study Director — University of Pennsylvania
Locations (7):
- United States (6):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No